CLINICAL TRIAL: NCT07199374
Title: PARCA (a Digital Tool) to Improve Justice and Health
Acronym: Parca
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: Q2i, LLC (Industry); RTI International (Other); Worcester Polytechnic Institute (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GeorgeMasonU; R42DA056255 (NIH)
Record Dates: First submitted 2025-03-19; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Behavioral Addiction
Keywords: probation supervision; recovery app

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PARCA App (Experimental): Officers and clients are using the application of PARCA which is on their phone and a web-based application. PARCA is a tool to detail goals and progress towards goals
  Interventions: Behavioral: PARCA
- Standard Supervision (No Intervention): Officers and clients are not using any new procedures or tools; they are using standard care.

INTERVENTIONS:
Behavioral: PARCA — PARCA is an s an app to facilitate goal management, resource allocation, and managing progress.
  Arms: PARCA App

SUMMARY:
The purpose of this study is to assess the effectiveness of the Probation/Parole and Reentry Coach Application (PARCA)-a mobile application that allows justice-involved people to set and manage personal goals to support sustained, successful community supervision. Through this study, we aim to conduct surveys and interviews aimed to gain a better understanding of ways to improve the substance use treatment process, connections between clients and officers, and goal selection and achievement for clients using the PARCA app

DETAILED DESCRIPTION:
This study tests a new technological intervention referred to as Probation/Parole and Reentry Coach Application (PARCA). The application uses motivational interviewing and cognitive behavioral techniques to engage clients in problem solving by identifying issues, identifying goals, making progress towards the goals, incentivizing clients to achieve the goals, and working towards completion of supervision. Officers can view the goals, progress, and points accumulated to improve supervision outcomes.

ELIGIBILITY:
Inclusion Criteria:

All officers that supervise individuals All individuals on supervision that indicate drug use -

Exclusion Criteria:

Individuals that have poor performance on their job clients have serious mental health disorders

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified gender
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of Days till the Individual Initiates Treatment | The timeframe is 365 days
  This represents the number of days that the individual starts treatment based on the day that they started supervision. This can be measured in the supervision records. This is an event in the record system like an electronic health record.

SECONDARY OUTCOMES:
Number of Treatment Sessions in 90 days | For 365 days
  This represents the number of times the individual participated in treatment during a 90 day window. This can be measured from supervision records.

OTHER OUTCOMES:
Drug Tests | through study completion, an average of 1 year
  Test positive for an illicit drug
Number of times the individual has been arrested or technically violated probation | This is for 365 days
  This criminal justice outcome refers to other criminal behavior and/or failure to abide by supervision conditions. Both reflect events that can be measured in the supervision records.

CONTACTS AND LOCATIONS:
Overall Officials: Faye S. Taxman, PhD, Principal Investigator — George Mason University
Locations (2):
- United States (2):
  - Travis County Community Services, Austin, Texas
  - Dallas County Community Supervision, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
These are confidential